CLINICAL TRIAL: NCT01118000
Title: Study on the Cardioprotection and Humoral Mechanism of Limb Ischemia Preconditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Guangdong Natural Science fund Committee, Guangdong Natural Science fund Committee
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDNSFC7001664
Record Dates: First submitted 2010-04-26; First posted 2010-05-06 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-04

CONDITIONS: Ischemic Preconditioning
Keywords: ischemic preconditioning,serum proteins,human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- limb ischemia preconditioning (Experimental): limb ischemic preconditioning consists of three 5-min cycles of left upper limb ischemia induced by a blood pressure cuff placed on the left upper arm and inflated to 200 mmHg,with an intervention 5-min of reperfusion during which the cuff was deflated.
  Interventions: Procedure: limb ischemia preconditioning

INTERVENTIONS:
Procedure: limb ischemia preconditioning — limb ischemic preconditioning consists of three 5-min cycles of left upper limb ischemia induced by a blood pressure cuff placed on the left upper arm and inflated to 200 mmHg,with an intervention 5-min of reperfusion during which the cuff was deflated.
  Other Names: remote ischemia preconditioning

SUMMARY:
Numerous studies Have shown that limb ischemic preconditioning can protect vital organs (including the heart) from ischemia-reperfusion injury,which has a broad application prospect.But its mechanism is still unclear. Evidence showed that humoral mechanisms may play an important role. This study was carried out on the limb ischemic preconditioning in healthy volunteers, collected their serum at different time points before and after treatment,classified and identified the serum proteins during different periods of limb ischemic preconditioning,by using methods including high abundant protein removal,Two-dimensional electrophoresis chromatography and mass spectrometry,then analysed activation and synthesis of the proteins in order to search for the proteins or peptides whose synthesis was activated by ischemic preconditioning. This study will be the first systemic explore of the changes in serum proteins of limb ischemic preconditioning in human body,and lay theoretical basis for the clinical application of limb ischemic preconditioning and for further explore of its humoral mechanism,thus provide clues for searching for protein or peptide having protective effects for organs.

DETAILED DESCRIPTION:
We aim to assess whether limb ischemic preconditioning protects remote tissue or organs through a humoral mechanism.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers aging 20-30 years old
* no cardiac，hepatic or renal，peripheral vascular diseases
* be willing to enter our study and sign an written informed consent

Exclusion Criteria:

* younger than 20 years old or older than 30 years old
* having cardiac，hepatic or renal，peripheral vascular diseases
* refuse to enter our study or sign an written informed consent

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Transient limb ischemia would change expression of several serum proteins in humans,indicating a humoral mechanism for its organ protection. | two years
  Proteomics analysis of the serum proteins.

SECONDARY OUTCOMES:
A questionnaire study of the acceptability of transient limb ischemia in healthy conscious subjects. | one year
  Transient limb ischemia as a remote ischemic preconditioning stimulus has been shown an effective and non-invasive strategy to protect remote tissue or organs from an extended ischemic event. But the acceptability of human subjects remains unknown. Our study aims to assess the acceptability of this transient limb ischemia protocol in healthy conscious subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jin S qing, Doctor, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- proteomics lab of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: PUMED — http://www.ncbi.nlm.nih.gov/sites/entrez
- See also: Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. — http://www.ncbi.nlm.nih.gov/pubmed/17707752
- See also: Ischemic preconditioning prevents endothelial injury and systemic neutrophil activation during ischemia-reperfusion in humans — http://www.ncbi.nlm.nih.gov/sites/entrez